CLINICAL TRIAL: NCT00323921
Title: Determination of Safety and Efficacy of a Laser With Cooling for Treatment of Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 052603
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Aged Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: dermatological infrared laser

SUMMARY:
The appearance of aged skin is a common cosmetic complaint of middle aged and older individuals. This study evaluates the safety and efficacy of a new laser with cooling to improve the appearance of aged skin. The laser being used will heat various depths of the skin while protecting the outer layer.

ELIGIBILITY:
Inclusion:

Aged skin, light to medium skin types.

Exclusion:

Known photosensitivity Any of the following pre-existing skin conditions: eczema, psoriasis, allergic dermatitis or other conditions that may affect treatment.

Other treatments within the past year for aged facial skin

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-08; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
score on a grading scale at post treatment visits

CONTACTS AND LOCATIONS:
Overall Officials: E. V. Ross, M.D., Principal Investigator — United States Naval Medical Center, San Diego